CLINICAL TRIAL: NCT01485770
Title: A Four-week, Double-blind, Placebo-controlled, Randomized, Cross-over Study of the Safety and Efficacy of ADX-N05 in the Treatment of Excessive Daytime Sleepiness
Brief Title: A Study of the Safety and Effectiveness of ADX-N05 in the Treatment of Excessive Daytime Sleepiness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ADX-N05 201
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Results first posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo, Then ADX-N05 (Experimental): Participants first receive a placebo to match ADX-N05 once a day for 2 consecutive weeks (Weeks 1 and 2). They will then receive ADX-N05 150 mg tablet once a day for seven days (Week 3) followed by 300 mg (2 tablets) once a day for seven days (Week 4).
  Interventions: Drug: ADX-N05; Drug: Placebo
- ADX-N05, Then Placebo (Placebo Comparator): Participants first receive ADX-N05 150 mg tablet once a day for seven days (Week 1) followed by 300 mg (2 tablets) once a day for seven days (Week 2). They will then receive a placebo to match ADX-N05 once a day for 2 consecutive weeks (Weeks 3 and 4).
  Interventions: Drug: ADX-N05; Drug: Placebo

INTERVENTIONS:
Drug: ADX-N05 — 150 mg once a day for seven days followed by 300 mg once a day for seven days
Drug: Placebo — Placebo to match ADX-N05 once a day for 2 consecutive weeks

SUMMARY:
This is a study to evaluate the safety and effectiveness of ADX-N05 compared to placebo in the treatment of excessive daytime sleepiness in adults with narcolepsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of narcolepsy
* Good general health
* Willing and able to comply with the study design and schedule and other requirements

Exclusion Criteria:

* If female, pregnant or lactating
* Customary bedtime later than midnight
* History of significant medical condition, behavioral or psychiatric disorder (including suicidal ideation), or surgical history
* Any other clinically relevant medical, behavioral or psychiatric disorder other than narcolepsy that is associated with excessive sleepiness
* History of significant cardiovascular disease
* Body mass index >34
* Excessive caffeine use - > 600 mg/day of caffeine or > 6 cups of coffee/day
* History of alcohol or drug abuse within the past two years
* Nicotine dependence that has an affect on sleep

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2011-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Pulmonary Associates, Phoenix, Arizona
  - Clinical Research Group of St. Petersburg, St. Petersburg, Florida
  - Neurotrials Research, Inc., Atlanta, Georgia
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - SleepMed of Central Georgia, Macon, Georgia
  - The Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - Mercy St. Anne Sleep Disorders Center, Toledo, Ohio
  - SleepMed of South Carolina, Columbia, South Carolina
  - Future Search Trials of Neurology, Austin, Texas
  - Sleep Medicine Associates of Texas, Dallas, Texas

REFERENCES:
- [Derived] Bogan RK, Feldman N, Emsellem HA, Rosenberg R, Lu Y, Bream G, Khayrallah M, Lankford DA. Effect of oral JZP-110 (ADX-N05) treatment on wakefulness and sleepiness in adults with narcolepsy. Sleep Med. 2015 Sep;16(9):1102-8. doi: 10.1016/j.sleep.2015.05.013. Epub 2015 Jun 3. PMID 26298786

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Then ADX-N05: Participants first received a placebo to match ADX-N05 once a day for 2 consecutive weeks (Weeks 1 and 2). They then received ADX-N05 150 mg tablet once a day for seven days (Week 3) followed by 300 mg (2 tablets) once a day for seven days (Week 4).
- ADX-N05, Then Placebo: Participants first received ADX-N05 150 mg tablet once a day for seven days (Week 1) followed by 300 mg (2 tablets) once a day for seven days (Week 2). They then received a placebo to match ADX-N05 once a day for 2 consecutive weeks (Weeks 3 and 4).
Period: First Intervention (2 Weeks)
Arm/Group | Placebo, Then ADX-N05 | ADX-N05, Then Placebo
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | Placebo, Then ADX-N05 | ADX-N05, Then Placebo
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, Then ADX-N05 | ADX-N05, Then Placebo | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.71 (11.56) | 42.81 (10.72) | 37.1 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 8 | 11 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 16 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Sleep Latency Time (in Minutes) as Determined From the Maintenance of Wakefulness Test (MWT) Following Two Weeks of Treatment With ADX-N05 vs. Two Weeks of Treatment With Placebo
Description: The MWT is a validated objective measure of the ability to stay awake for a defined period of time. The change from baseline in the mean sleep latency from the MWT was the average of sleep latency from the four trials of the MWT.
Time Frame: Baseline up to 2 weeks post-dose.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- ADX-N05 300 mg: Participants took 2 tablets of 150 mg (300 mg) ADX-N05 once a day during week 2 or week 4 of the 4-week study treatment period.
- Placebo: Participants took Placebo to match ADX-N05 once a day during week 2 or week 4 of the 4-week study treatment period.
Arm/Group | ADX-N05 300 mg | Placebo
Number analyzed (Participants) | 33 | 33
minutes | 12.7 (10.64) | 0.9 (6.02)

2. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Score During Weeks 1 and 3
Description: The ESS is a questionnaire intended to measure daytime sleepiness. In this test, participants answer questions with regard to the level of sleepiness they experienced over approximately the 7 days prior to the assessment while performing eight common, non-stimulating activities. The ESS total score range is 1 to 24. Each activity is rated on a 4-point scale ranging from a minimum of "would never doze" to a maximum of "a high chance of dozing." Thus, the ESS scale range is as follows: 0=would never doze, 1=slight chance of dozing, 2=moderate chance of dozing, 3=high chance of dozing; 0 indicates a better outcome, and 3 indicates a worse outcome. A negative mean change value indicates a decrease in score from baseline and an improvement in daytime sleepiness.
Time Frame: Baseline up to Week 3 post-dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- ADX-N05 150 mg: Participants took 1 tablet of 150 mg ADX-N05 once a day during week 1 or week 3 of the 4-week study treatment period.
- Placebo: Participants took Placebo to match ADX-N05 once a day during week 1 or week 3 of the 4-week study treatment period.
Arm/Group | ADX-N05 150 mg | Placebo
Number analyzed (Participants) | 33 | 33
score on a scale | -5.3 (5.20) | -1.2 (4.09)

3. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Score During Weeks 2 and 4
Description: as for outcome 2
Time Frame: Baseline up to Week 4 post-dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ADX-N05 300 mg | Placebo
Number analyzed (Participants) | 33 | 33
score on a scale | -6.7 (6.15) | -2.4 (3.82)

4. Secondary Outcome: Number of Participants With Improved Clinical Global Impression of Change (CGI-C) Scores During Weeks 1 and 3
Description: The CGI-C scale was completed at Week 1 through 4 visits. The participant was rated on a 7-point scale ranging from a minimum of "Very much improved" to a maximum of "Very much worse." The proportion of participants experiencing at least minimal improvement on the CGI-C was calculated and summarized for each of the two weeks of each of the treatment periods. The CGI-C scale consists of the following ratings: 1-Very Much improved, 2-Much improved, 3-Minimally improved, 4-No change, 5-Minimally worse, 6-Much worse, 7-Very much worse; a rating of 1 indicates a better outcome, and a rating of 7 indicates a worse outcome. Improvement was defined as a CGI-rating of 1, 2, or 3.
Time Frame: Week 1 and Week 3 post-dose.
Measure: Count of Participants; unit: Participants
Arm/Group | ADX-N05 150 mg | Placebo
Number analyzed (Participants) | 33 | 33
Participants | 29 | 9

5. Secondary Outcome: Number of Participants With Improved Clinical Global Impression of Change (CGI-C) Scores During Weeks 2 and 4
Description: as for outcome 4
Time Frame: Week 2 and Week 4 post-dose.
Measure: Count of Participants; unit: Participants
Arm/Group | ADX-N05 300 mg | Placebo
Number analyzed (Participants) | 33 | 33
Participants | 25 | 13

ADVERSE EVENTS:
Groups:
- ADX-N05: Participants received ADX-N05 150 mg once a day for seven days followed by 300 mg once a day for seven days during the 4-week study treatment period.
- Placebo: Participants received Placebo to match ADX-N05 once a day for 2 consecutive weeks during the 4-week study treatment period.
Arm/Group | ADX-N05 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 20/33 | 0/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADX-N05 (N=33) | Placebo (N=33)
Headache (Nervous system disorders) | 3 | 0
Initial Insomnia (Nervous system disorders) | 2 | 0
Insomnia (Nervous system disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 0
Chest discomfort (General disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 2 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No